CLINICAL TRIAL: NCT01067261
Title: Transcutaneous Mechanical Nerve Stimulation (TMNS) by Vibration in the Preservation and Restoration of Urinary Continence and Erectile Function and in the Treatment of Erectile Dysfunction and Urinary Incontinence in Conjunction With Nerve Sparing Radical Prostatectomy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Copenhagen University Hospital at Herlev (Other)
Collaborators: Aarhus University Hospital Skejby (Other); Velux Fonden (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HC-2008-127
Record Dates: First submitted 2010-02-10; First posted 2010-02-11 (Estimated); Last update posted 2013-05-24 (Estimated); Status verified 2012-12

CONDITIONS: Erectile Dysfunction; Urinary Incontinence
Keywords: Nerve stimulation; TMNS; Prostatectomy; Prevention; Restoration; Treatment; Vibration; Non-invasive
MeSH Terms: conditions — Erectile Dysfunction; Urinary Incontinence

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- TMNS and pelvic floor muscle training (Experimental): This group will receive both the normal pelvic floor muscle training and the TMNS vibration therapy following their radical prostatectomy. Treatment with TMNS will start before the surgery and continue 6 weeks after the surgery.
  Interventions: Device: Transcutaneous mechanical nerve stimulation (TMNS)
- Pelvic floor muscle training only (Active Comparator): This group will receive the normal pelvic floor muscle training after prostatectomy only.
  Interventions: Other: Pelvic floor muscle training

INTERVENTIONS:
Device: Transcutaneous mechanical nerve stimulation (TMNS) — Device: Transcutaneous mechanical nerve stimulation by A medical vibrator (FERTI CARE personel, Multicept A/S, Albertslund, Danmark)
  A medical vibrator (FERTI CARE personel, Multicept A/S, Albertslund, Denmark) will be used. The stimulation works through a vibrating disc of hard plastic with a diameter of 3.5 cm. The stimulation point will be the frenulum. A stimulation sequence consisting of 10 seconds of stimulation followed by a 10 second pause repeated 10 times will be used. The treatment will be initiated 1 to 4 weeks before the radical prostatectomy and re-initiated 0 to 14 days after the operation. The treatment will then continue for 6 weeks. The stimulation will be preformed daily by the patients in their own homes.
  Other Names: FERTI CARE personel, Multicept A/S, Albertslund, Danmark
  Arms: TMNS and pelvic floor muscle training
Other: Pelvic floor muscle training — Regular pelvic floor training which is offered to all patients undergoing a radical prostatectomy at Herlev Hospital.
  Arms: Pelvic floor muscle training only

SUMMARY:
After radical prostatectomy nerve damage in the pelvic floor usually occurs. This causes side effects in the form of incontinence and erectile dysfunction.

It has previously been shown that one can stimulate the nerves of the pelvic floor by means of transcutaneous mechanical nerve stimulation (TMNS) done through vibration. This study will examine the effect of TMNS in the preservation and restoration of urinary continence and erectile function and in the treatment of urinary incontinence and erectile dysfunction in conjunction with radical prostatectomy.

The theory is that by means of TMNS one can stimulate the nerves of the pelvic floor and the penis which may improve their function and there by prevent or minimize the occurrence of incontinence and erectile dysfunction following pelvic surgery. Vibration may also help to eliminate these symptoms once they have occurred. It is possible that TMNS will also directly increase the blood flow in the cavernosal tissue thus aiding in the preservation of this tissue. In case the improved nerve function is not great enough to secure satisfactory erectile function in itself it may still improve the effect of PDE-5-inhibitors.

In pilot studies TMNS has already shown an effect in the treatment of urinary continence.

In this study the patients will be randomized to either TMNS treatment or no TMNS treatment. In both groups the patients will participate in a pelvic floor muscle training program. In the group receiving active treatment this will be supplemented by TMNS treatment. The two groups will be evaluated and compared with regard to erectile function time to continence after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled to undergo nerve sparing radical prostatectomy
* Continent before surgery
* A minimum score on the IIEF-questionnaire of 18
* Sexually active

Exclusion Criteria:

* Treatment with nitrates
* Treatment with α-blockers
* Serious cardiovascular disease
* Severely reduced liver function,
* Retinitis pigmentosa,
* Non-arteritic ischemic optic neuropathy (NAION)
* Previous vascular infarction of the eye

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2010-02; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Erectile function score by a validated symptom questionnaire (IIEF) | At 3 months, 6 months and 1 year
Time to continence after surgery | At 3 months, 6 months and 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Jens R Sønksen, MD, Ph.D, Study Director — Copenhagen University Hospital at Herlev
Locations (2):
- Denmark (2):
  - Department of Urology, Aarhus University Hospital, Skejby, Aarhus N
  - Department of Urology, Herlev University Hospital, Herlev

REFERENCES:
- [Derived] Fode M, Borre M, Ohl DA, Lichtbach J, Sonksen J. Penile vibratory stimulation in the recovery of urinary continence and erectile function after nerve-sparing radical prostatectomy: a randomized, controlled trial. BJU Int. 2014 Jul;114(1):111-7. doi: 10.1111/bju.12501. Epub 2014 Jan 22. PMID 24127838